CLINICAL TRIAL: NCT02051907
Title: A BLIND, CONTROLLED CLINICAL STUDY TO EVALUATE THE EFFICACY AND SAFETY OF KAM1403 GEL TREATMENT IN PATIENTS WITH RADIATION DERMATITIS
Brief Title: Clinical Study to Evaluate Safety and Efficacy of KAM1403 Gel to Treat Radiation Dermatitis
Acronym: kam1403
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kamedis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAM-RAD-01
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- KAM1403 Gel (Experimental): A group treated with KAM1403 for the study period.
  Interventions: Device: KAM1403 Gel
- Aloevera Gel (Sham Comparator): A group treated with Aloevera Gel for the study period
  Interventions: Device: aloevera gel

INTERVENTIONS:
Device: KAM1403 Gel
  Arms: KAM1403 Gel
Device: aloevera gel
  Arms: Aloevera Gel

SUMMARY:
The main purpose of this study is to demonstrate the safety and efficacy of KAM1403 GEL in reducing the symptoms of mild to moderate Radiation Dermatitis. Efficacy will be evaluated by comparing symptoms assessment during and post radiotherapy: erythema, desquamation, edema, moist desquamation and ulceration in the KAM1403 Gel treated group versus a group of subjects treated with the Aloe vera Gel (the control group). In addition, a comparison will be made between subjects' self evaluation in the treatment group versus the control group. Safety will be determined by the number and severity of Adverse Events Device-Related.

ELIGIBILITY:
Inclusion Criteria:

* Female above 18 years of age
* Diagnosed with breast cancer and scheduled to receive postoperative radiotherapy
* Treatment of regional lymph nodes (i.e. axillary, supraclavicular, or internal mammary) is allowed.
* Schedule for breast radiotherapy (RT) to a dose of 50 Gy in 2 Gy/fx, for 5 weeks and then a boost to the lumpectomy cavity.
* Minimum of 3 weeks from chemotherapy to start of radiation therapy.
* Patient agrees to use only the test products during the study period

Exclusion Criteria:

* Tumor involvement of the skin
* Patient has another dermatological disease/condition that could interfere with clinical evaluation including infected atopic dermatitis lesions
* Patient has a previous history of allergy to the ingredients of the tested formulations
* Paget's disease of the nipple.
* Pregnant or lactating females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Radiation dermatitis symptoms | Day 0, weeks 2, 4, 6.5, 8.5
  Changes in Radiation dermatitis symptoms assessment during and post radiotherapy (erythema, desquamation, edema, moist desquamation and ulceration) using the Radiation Therapy Oncology Group toxicity scoring system in the treatment group versus the control group

SECONDARY OUTCOMES:
Subjects' self evaluation | Day 0, weeks 2, 4, 6.5, 8.5
Number of Adverse Events | Day 0, weeks 2, 4, 6.5, 8.5

CONTACTS AND LOCATIONS:
Overall Officials: Diana Matchiavsky, MD, Principal Investigator — Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- See also: Sponsor's site — http://www.kamedis.com